CLINICAL TRIAL: NCT02693548
Title: The Spanish Familial Hypercholesterolaemia Cohort Study
Acronym: SAFEHEART
Status: Recruiting | Type: Observational
Sponsor: Fundación Hipercolesterolemia Familiar (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Fundación Centro Nacional de Investigaciones Cardiovasculares Carlos III (Other)
Responsible Party: Sponsor
Other Study IDs: SAFEHEART
Record Dates: First submitted 2016-02-09; First posted 2016-02-26 (Estimated); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Familial Hypercholesterolaemia
Keywords: Familial Hypercholesterolaemia; Prognosis; Cardiovascular disease
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples were taken after 12 hours of fasting. Serum, plasma and DNA samples were aliquoted and preserved at -80°C. Serum total cholesterol, triglycerides and HDL-cholesterol levels were measured in a centralized laboratory using enzymatic methods
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Familial hypercholesterolaemia patients: Index cases with genetic diagnosis of FH and their relatives over 15 years old with a genetic diagnosis of FH.
- Unaffected relatives: Relatives of FH patients without FH (genetically defined)

SUMMARY:
SAFEHEART is a large, on-going registry study in molecularly defined patients with heterozygous FH treated in Spain.

DETAILED DESCRIPTION:
Familiar hypercholesterolemia (FH) is the most common genetic disorder associated with the development of severe and premature coronary artery disease (CAD). The disorder is caused by mutations in the gene that encodes the low-density lipoprotein receptor (LDL-r), resulting in a lower expression of functional LDL-r in the liver. FH has autosomal dominant transmission with high penetrance and the prevalence of heterozygous individuals is one in 400 to 500 in the general population. To date, more than 800 different functional mutations of the LDL-r gene have been described worldwide, and more than 200 have been documented in Spain. In addition, a much less common disorder that resemble FH is familial defective apoB 100 disorder (FDB) produced by a mutation in the Apo B 100 gene. FDB accounts for a significant proportion of FH in some localized regions of Spain.

Life expectancy is shortened by 20 to 30 years in FH patients, and sudden death and myocardial infarction are the principal causes of death. The Simon Broome Register of FH in Great Britain, has shown that FH has a 100-fold increase in coronary mortality and a nearly 10-fold increase in total mortality, especially in young adults.

Since the 1990's, coronary mortality and total mortality in FH patients have decreased remarkably in part due to the use of more effective lipid-lowering therapy such as statins. The analysis of the Dutch FH cohort showed that an early treatment with statins after the diagnosis of the disorder leads to near normalisation of coronary heart disease risk comparable to the general population. Therefore, most of patients require an early, continuous and more intensive lipid-lowering therapy.

Despite the use of statins, this population still have a high risk for the development of premature CAD. Therefore, the need to study the relatives of a known FH case, know as cascade screening, is essential to detect those cases that are younger, probably with a less severe form of FH and are not receiving treatment to prevent cardiovascular disease development.

Although the genetic defect is probably the most important factor in the clinical expression of FH, other genetic (gene-gene interactions), environmental (particularly those relating to diet, tobacco consumption and physical activity) and metabolic factors could play an important role in modulating the atherosclerotic burden in this population.

To gain insight into the prognostic factors and mechanisms that influence the development of CAD and mortality in FH, a long-term prospective follow-up of a molecularly well-defined FH cohort using a multidisciplinary approach is necessary. This cohort is an excellent tool of translational research to evaluate and determine the principal prognostic factors related to CAD morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Index cases with genetic diagnosis of FH and their relatives over 15 years old with a genetic diagnosis of FH and their first-degree relatives

Exclusion Criteria:

* Patient unwillingness

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Index cases with genetic diagnosis of FH and their relatives over 15 years old with a genetic diagnosis of FH and their unaffected relatives
Sampling Method: Non-Probability Sample
Enrollment: 4141 (Estimated)
Dates: Start 2004-01 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Prognostic assessment: time to fatal or non-fatal cardiovascular event. | up to 12 years
  Time to first cardiovascular event: fatal or non-fatal myocardial infarction, fatal or non-fatal ischemic stroke, coronary revascularization, peripheral artery revascularization, aortic valve replacement or cardiovascular death.

SECONDARY OUTCOMES:
LDL-cholesterol level (mg/dl) at entry and at follow-up | up to12 years
  LDL-cholesterol measurement at enrolment and after follow-up. At enrolment, a central core lab is in charge of the analysis. During follow-up, a yearly-based phone call is used to contact every subject and a complete lipid profile is obtained from the patient (obtained in his/her usual medical care).

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Mata, MD, Study Chair — Fundacion Hipercolesterolemia Familiar
Locations (1):
- Fundacion Hipercolesterolemia Familiar, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Available access for publication

REFERENCES:
- [Background] Vallejo-Vaz AJ, Kondapally Seshasai SR, Cole D, Hovingh GK, Kastelein JJ, Mata P, Raal FJ, Santos RD, Soran H, Watts GF, Abifadel M, Aguilar-Salinas CA, Akram A, Alnouri F, Alonso R, Al-Rasadi K, Banach M, Bogsrud MP, Bourbon M, Bruckert E, Car J, Corral P, Descamps O, Dieplinger H, Durst R, Freiberger T, Gaspar IM, Genest J, Harada-Shiba M, Jiang L, Kayikcioglu M, Lam CS, Latkovskis G, Laufs U, Liberopoulos E, Nilsson L, Nordestgaard BG, O'Donoghue JM, Sahebkar A, Schunkert H, Shehab A, Stoll M, Su TC, Susekov A, Widen E, Catapano AL, Ray KK. Familial hypercholesterolaemia: A global call to arms. Atherosclerosis. 2015 Nov;243(1):257-9. doi: 10.1016/j.atherosclerosis.2015.09.021. Epub 2015 Sep 18. No abstract available. PMID 26408930
- [Background] Fuentes F, Alcala-Diaz JF, Watts GF, Alonso R, Muniz O, Diaz-Diaz JL, Mata N, Sanchez Munoz-Torrero JF, Brea A, Galiana J, Figueras R, Aguado R, Piedecausa M, Cepeda JM, Vidal JI, Rodriguez-Cantalejo F, Lopez-Miranda J, Mata P; SAFEHEART Investigators. Statins do not increase the risk of developing type 2 diabetes in familial hypercholesterolemia: The SAFEHEART study. Int J Cardiol. 2015 Dec 15;201:79-84. doi: 10.1016/j.ijcard.2015.07.107. Epub 2015 Aug 5. PMID 26296047
- [Background] Alonso R, Andres E, Mata N, Fuentes-Jimenez F, Badimon L, Lopez-Miranda J, Padro T, Muniz O, Diaz-Diaz JL, Mauri M, Ordovas JM, Mata P; SAFEHEART Investigators. Lipoprotein(a) levels in familial hypercholesterolemia: an important predictor of cardiovascular disease independent of the type of LDL receptor mutation. J Am Coll Cardiol. 2014 May 20;63(19):1982-9. doi: 10.1016/j.jacc.2014.01.063. Epub 2014 Mar 13. PMID 24632281
- [Background] Alonso R, Mata P, Zambon D, Mata N, Fuentes-Jimenez F. Early diagnosis and treatment of familial hypercholesterolemia: improving patient outcomes. Expert Rev Cardiovasc Ther. 2013 Mar;11(3):327-42. doi: 10.1586/erc.13.7. PMID 23469913
- [Background] Aledo R, Alonso R, Mata P, Llorente-Cortes V, Padro T, Badimon L. LRP1 gene polymorphisms are associated with premature risk of cardiovascular disease in patients with familial hypercholesterolemia. Rev Esp Cardiol (Engl Ed). 2012 Sep;65(9):807-12. doi: 10.1016/j.recesp.2012.03.013. Epub 2012 Jul 20. English, Spanish. PMID 22819221
- [Background] Vazquez C, Alonso R, Garriga M, de Cos A, de la Cruz JJ, Fuentes-Jimenez F, Salas-Salvado J, Mata P. Validation of a food frequency questionnaire in Spanish patients with familial hypercholesterolaemia. Nutr Metab Cardiovasc Dis. 2012 Oct;22(10):836-42. doi: 10.1016/j.numecd.2011.01.007. Epub 2011 Jun 23. PMID 21703832
- [Background] Mata N, Alonso R, Badimon L, Padro T, Fuentes F, Muniz O, Perez-Jimenez F, Lopez-Miranda J, Diaz JL, Vidal JI, Barba A, Piedecausa M, Sanchez JF, Irigoyen L, Guallar E, Ordovas JM, Mata P. Clinical characteristics and evaluation of LDL-cholesterol treatment of the Spanish Familial Hypercholesterolemia Longitudinal Cohort Study (SAFEHEART). Lipids Health Dis. 2011 Jun 10;10:94. doi: 10.1186/1476-511X-10-94. PMID 21663647
- [Background] Criado-Garcia J, Fuentes F, Cruz-Teno C, Garcia-Rios A, Jimenez-Morales A, Delgado-Lista J, Mata P, Alonso R, Lopez-Miranda J, Perez-Jimenez F; Spanish Group for the Study of Familiar Hypercholesterolemia. R353Q polymorphism in the factor VII gene and cardiovascular risk in Heterozygous Familial Hypercholesterolemia: a case-control study. Lipids Health Dis. 2011 Apr 9;10:50. doi: 10.1186/1476-511X-10-50. PMID 21477332
- [Background] Garcia-Rios A, Perez-Martinez P, Mata P, Fuentes F, Lopez-Miranda J, Alonso R, Caballero J, Mata N, Perez-Jimenez F, Ordovas JM. Polymorphism at the TRIB1 gene modulates plasma lipid levels: insight from the Spanish familial hypercholesterolemia cohort study. Nutr Metab Cardiovasc Dis. 2011 Dec;21(12):957-63. doi: 10.1016/j.numecd.2010.04.002. Epub 2010 Aug 6. PMID 20692138
- [Background] Zambon D, Quintana M, Mata P, Alonso R, Benavent J, Cruz-Sanchez F, Gich J, Pocovi M, Civeira F, Capurro S, Bachman D, Sambamurti K, Nicholas J, Pappolla MA. Higher incidence of mild cognitive impairment in familial hypercholesterolemia. Am J Med. 2010 Mar;123(3):267-74. doi: 10.1016/j.amjmed.2009.08.015. PMID 20193836
- [Background] Garcia-Rios A, Perez-Martinez P, Fuentes F, Mata P, Lopez-Miranda J, Alonso R, Rodriguez F, Garcia-Olid A, Ruano J, Ordovas JM, Perez-Jimenez F. Genetic variations at ABCG5/G8 genes modulate plasma lipids concentrations in patients with familial hypercholesterolemia. Atherosclerosis. 2010 Jun;210(2):486-92. doi: 10.1016/j.atherosclerosis.2010.01.010. Epub 2010 Jan 22. PMID 20172523
- [Background] Alonso R, Defesche JC, Tejedor D, Castillo S, Stef M, Mata N, Gomez-Enterria P, Martinez-Faedo C, Forga L, Mata P. Genetic diagnosis of familial hypercholesterolemia using a DNA-array based platform. Clin Biochem. 2009 Jun;42(9):899-903. doi: 10.1016/j.clinbiochem.2009.01.017. Epub 2009 Feb 6. PMID 19318025
- [Background] Alonso R, Mata N, Castillo S, Fuentes F, Saenz P, Muniz O, Galiana J, Figueras R, Diaz JL, Gomez-Enterria P, Mauri M, Piedecausa M, Irigoyen L, Aguado R, Mata P; Spanish Familial Hypercholesterolaemia Group. Cardiovascular disease in familial hypercholesterolaemia: influence of low-density lipoprotein receptor mutation type and classic risk factors. Atherosclerosis. 2008 Oct;200(2):315-21. doi: 10.1016/j.atherosclerosis.2007.12.024. Epub 2008 Feb 20. PMID 18243212
- [Background] Merino-Ibarra E, Castillo S, Mozas P, Cenarro A, Martorell E, Diaz JL, Suarez-Tembra M, Alonso R, Civeira F, Mata P, Pocovi M; Spanish Group of Familial Hypercholesterolemia. Screening of APOB gene mutations in subjects with clinical diagnosis of familial hypercholesterolemia. Hum Biol. 2005 Oct;77(5):663-73. PMID 16596945
- [Background] Civeira F, Castillo S, Alonso R, Merino-Ibarra E, Cenarro A, Artied M, Martin-Fuentes P, Ros E, Pocovi M, Mata P; Spanish Familial Hypercholesterolemia Group. Tendon xanthomas in familial hypercholesterolemia are associated with cardiovascular risk independently of the low-density lipoprotein receptor gene mutation. Arterioscler Thromb Vasc Biol. 2005 Sep;25(9):1960-5. doi: 10.1161/01.ATV.0000177811.14176.2b. Epub 2005 Jul 14. PMID 16020744
- [Background] Alonso R, Castillo S, Civeira F, Puzo J, de la Cruz JJ, Pocovi M, Mata P. [Heterozygous familial hypercholesterolemia in Spain. Description of 819 non related cases]. Med Clin (Barc). 2002 Apr 13;118(13):487-92. doi: 10.1016/s0025-7753(02)72428-7. Spanish. PMID 11975885
- [Background] Castillo S, Tejedor D, Mozas P, Reyes G, Civeira F, Alonso R, Ros E, Pocovi M, Mata P. The apolipoprotein B R3500Q gene mutation in Spanish subjects with a clinical diagnosis of familial hypercholesterolemia. Atherosclerosis. 2002 Nov;165(1):127-35. doi: 10.1016/s0021-9150(02)00190-9. PMID 12208478
- [Background] Alonso R, Mata P, De Andres R, Villacastin BP, Martinez-Gonzalez J, Badimon L. Sustained long-term improvement of arterial endothelial function in heterozygous familial hypercholesterolemia patients treated with simvastatin. Atherosclerosis. 2001 Aug;157(2):423-9. doi: 10.1016/s0021-9150(00)00733-4. PMID 11472743
- [Derived] de Isla LP, Vallejo-Vaz AJ, Watts GF, Muniz-Grijalvo O, Alonso R, Diaz-Diaz JL, Arroyo-Olivares R, Aguado R, Argueso R, Mauri M, Romero MJ, Alvarez-Banos P, Manas D, Cepeda JM, Gonzalez-Bustos P, Casanas M, Michan A, Munoz-Torrero JFS, Faedo C, Barba MA, Dieguez M, de Andres R, Hernandez AM, Gonzalez-Estrada A, Padro T, Fuentes F, Badimon L, Mata P; SAFEHEART Investigators. Long-term sex differences in atherosclerotic cardiovascular disease in individuals with heterozygous familial hypercholesterolaemia in Spain: a study using data from SAFEHEART, a nationwide, multicentre, prospective cohort study. Lancet Diabetes Endocrinol. 2024 Sep;12(9):643-652. doi: 10.1016/S2213-8587(24)00192-X. Epub 2024 Aug 1. PMID 39098315
- [Derived] Alonso R, Arroyo-Olivares R, Diaz-Diaz JL, Fuentes-Jimenez F, Arrieta F, de Andres R, Gonzalez-Bustos P, Argueso R, Martin-Ordiales M, Martinez-Faedo C, Illan F, Saenz P, Donate JM, Sanchez Munoz-Torrero JF, Martinez-Hervas S, Mata P. Improved lipid-lowering treatment and reduction in cardiovascular disease burden in homozygous familial hypercholesterolemia: The SAFEHEART follow-up study. Atherosclerosis. 2024 Jun;393:117516. doi: 10.1016/j.atherosclerosis.2024.117516. Epub 2024 Mar 16. PMID 38523000
- [Derived] Alonso R, Arroyo-Olivares R, Muniz-Grijalvo O, Diaz-Diaz JL, Munoz-Torrero JS, Romero MJ, de Andres R, Zambon D, Manas MD, Fuentes-Jimenez F, Aguado R, Alvarez-Banos P, Arrieta F, Gonzalez-Bustos P, Cepeda J, Martin-Ordiales M, Mosquera D, Michan A, de Isla LP, Argueso R, Mata P. Persistence with long-term PCSK9 inhibitor treatment and its effectiveness in familial hypercholesterolaemia: data from the SAFEHEART study. Eur J Prev Cardiol. 2023 Mar 1;30(4):320-328. doi: 10.1093/eurjpc/zwac277. PMID 36416136
- [Derived] Perez de Isla L, Watts GF, Muniz-Grijalvo O, Diaz-Diaz JL, Alonso R, Zambon D, Fuentes-Jimenez F, Mauri M, Padro T, Vidal-Pardo JI, Barba MA, Ruiz-Perez E, Michan A, Mediavilla JD, Hernandez AM, Romero-Jimenez MJ, Badimon L, Mata P; SAFEHEART Investigators. A resilient type of familial hypercholesterolaemia: case-control follow-up of genetically characterized older patients in the SAFEHEART cohort. Eur J Prev Cardiol. 2022 May 5;29(5):795-801. doi: 10.1093/eurjpc/zwab185. PMID 34864959
- [Derived] Perez de Isla L, Watts GF, Alonso R, Diaz-Diaz JL, Muniz-Grijalvo O, Zambon D, Fuentes F, de Andres R, Padro T, Lopez-Miranda J, Mata P. Lipoprotein(a), LDL-cholesterol, and hypertension: predictors of the need for aortic valve replacement in familial hypercholesterolaemia. Eur Heart J. 2021 Jun 7;42(22):2201-2211. doi: 10.1093/eurheartj/ehaa1066. PMID 33437997
- [Derived] Perez de Isla L, Alonso R, Gomez de Diego JJ, Muniz-Grijalvo O, Diaz-Diaz JL, Zambon D, Miramontes JP, Fuentes F, de Andres R, Werenitzky J, Padro T, Saltijeral A, Mata P; SAFEHEART investigators. Coronary plaque burden, plaque characterization and their prognostic implications in familial hypercholesterolemia: A computed tomographic angiography study. Atherosclerosis. 2021 Jan;317:52-58. doi: 10.1016/j.atherosclerosis.2020.11.012. Epub 2020 Nov 18. PMID 33261814
- [Derived] Perez de Isla L, Arroyo-Olivares R, Alonso R, Muniz-Grijalvo O, Diaz-Diaz JL, Zambon D, Fuentes F, Mata N, Piedecausa M, Manas MD, Sanchez Munoz-Torrero JF, Miramontes-Gonzalez JP, de Andres R, Mauri M, Aguado R, Brea A, Cepeda JM, Vidal-Pardo JI, Martinez-Faedo C, Barba MA, Argueso R, Ruiz-Perez E, Michan A, Arrieta F, Riestra Fernandez M, Perez L, Pinilla JM, Diaz-Soto G, Pinto X, Padro T, Badimon L, Mata P; SAFEHEART researchers. Incidence of cardiovascular events and changes in the estimated risk and treatment of familial hypercholesterolemia: the SAFEHEART registry. Rev Esp Cardiol (Engl Ed). 2020 Oct;73(10):828-834. doi: 10.1016/j.rec.2019.10.028. Epub 2020 Mar 20. English, Spanish. PMID 32201274
- [Derived] Perez de Isla L, Alonso R, Muniz-Grijalvo O, Diaz-Diaz JL, Zambon D, Miramontes JP, Fuentes F, Gomez de Diego JJ, Gonzalez-Estrada A, Mata N, Saltijeral A, Barreiro M, Tomas M, de Andres R, Argueso R, Serrano Gotarredona MP, Navarro Herrero S, Perea Palazon RJ, de Caralt TM, Suarez de Centi LA, Zhilina S, Espejo Perez S, Padro T, Mata P; SAFEHEART investigators. Coronary computed tomographic angiography findings and their therapeutic implications in asymptomatic patients with familial hypercholesterolemia. Lessons from the SAFEHEART study. J Clin Lipidol. 2018 Jul-Aug;12(4):948-957. doi: 10.1016/j.jacl.2018.04.003. Epub 2018 Apr 17. PMID 29753733
- [Derived] Lazaro P, Perez de Isla L, Watts GF, Alonso R, Norman R, Muniz O, Fuentes F, Mata N, Lopez-Miranda J, Gonzalez-Juanatey JR, Diaz-Diaz JL, Blasco AJ, Mata P. Cost-effectiveness of a cascade screening program for the early detection of familial hypercholesterolemia. J Clin Lipidol. 2017 Jan-Feb;11(1):260-271. doi: 10.1016/j.jacl.2017.01.002. Epub 2017 Jan 10. PMID 28391894
- [Derived] Perez de Isla L, Alonso R, Mata N, Fernandez-Perez C, Muniz O, Diaz-Diaz JL, Saltijeral A, Fuentes-Jimenez F, de Andres R, Zambon D, Piedecausa M, Cepeda JM, Mauri M, Galiana J, Brea A, Sanchez Munoz-Torrero JF, Padro T, Argueso R, Miramontes-Gonzalez JP, Badimon L, Santos RD, Watts GF, Mata P. Predicting Cardiovascular Events in Familial Hypercholesterolemia: The SAFEHEART Registry (Spanish Familial Hypercholesterolemia Cohort Study). Circulation. 2017 May 30;135(22):2133-2144. doi: 10.1161/CIRCULATIONAHA.116.024541. Epub 2017 Mar 8. PMID 28275165
- [Derived] Perez de Isla L, Alonso R, Mata N, Saltijeral A, Muniz O, Rubio-Marin P, Diaz-Diaz JL, Fuentes F, de Andres R, Zambon D, Galiana J, Piedecausa M, Aguado R, Mosquera D, Vidal JI, Ruiz E, Manjon L, Mauri M, Padro T, Miramontes JP, Mata P; SAFEHEART Investigators. Coronary Heart Disease, Peripheral Arterial Disease, and Stroke in Familial Hypercholesterolaemia: Insights From the SAFEHEART Registry (Spanish Familial Hypercholesterolaemia Cohort Study). Arterioscler Thromb Vasc Biol. 2016 Sep;36(9):2004-10. doi: 10.1161/ATVBAHA.116.307514. Epub 2016 Jul 21. PMID 27444203